CLINICAL TRIAL: NCT06415045
Title: The Effect of Food on the Pharmacokinetics of BI 1015550 (Formulation C2) Following Single Oral Dose Administration in Healthy Subjects (an Open-label, Randomised, Single-dose, Two-period, Two-sequence Crossover Design)
Brief Title: A Study in Healthy People to Test How BI 1015550 is Taken up in the Body When Given With or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0039; 2023-509889-38-00 (Registry Identifier: CTIS); U1111-1301-0891 (Other: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerandomilast fasted state (Reference (R))/Nerandomilast fed state Test (T) (Experimental): Nerandomilast fasted state Reference (R)/Nerandomilast fed state Test (T)
  Two period crossover separated by a wash-out of at least 10 days:
  Period 1: Participants received one 18 mg Nerandomilast Formulation C2 film-coated tablet following an overnight fast of at least 10 hours.
  Period 2: Participants received One 18 mg Nerandomilast Formulation C2 film-coated tablet following a high fat/high calorie meal.
  Interventions: Drug: BI 1015550
- Nerandomilast fed state (Test (T))/Nerandomilast fasted state (Reference (R)) (Experimental): Nerandomilast fed state Test (T)/Nerandomilast fasted state Reference (R)
  Two period crossover separated by a wash-out of at least 10 days:
  Period 1: Participants received One 18 mg Nerandomilast Formulation C2 film-coated tablet following a high fat/high calorie meal.
  Period 2: Participants received one 18 mg Nerandomilast Formulation C2 film-coated tablet following an overnight fast of at least 10 hours.
  Interventions: Drug: BI 1015550

INTERVENTIONS:
Drug: BI 1015550 — Participants received a single 18 mg Nerandomilast Formulation C2 film-coated tablet either after an overnight fast of at least 10 hours or following a high-fat, high-calorie meal.
  Other Names: Nerandomilast; JASCAYD®

SUMMARY:
The main objective is to investigate the effect of food on the pharmacokinetics of BI 1015550 Formulation C2.

ELIGIBILITY:
Inclusion Criteria :

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m^2 (inclusive)
* Signed and dated written informed consent in accordance with International Conference of Harmonization-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Female subject who meets the criteria defined in the protocol for a highly effective contraception from at least 30 days before the first administration of trial medication until 7 days after last administration

Exclusion Criteria :

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 betas per minute (bpm) at screening
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, in particular, hepatic parameters (Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), total bilirubin) or renal parameters (creatinine) exceeding the upper limit of normal (ULN) at screening
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders assessed as clinically relevant by the investigator
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders including but not limited to depression and suicidal behavior
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label, single-dose, 2-period, 2-sequence crossover trial investigated how food affects the pharmacokinetics of an 18 mg nerandomilast tablet (Formulation C2). Subjects received nerandomilast in a fasting (Reference (R)) and fed (Test (T)) state with a minimum 10-day washout period in between and were randomized to the sequences R-T or T-R.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: period 1
Arm/Group | Nerandomilast fasted state (Reference (R))/Nerandomilast fed state Test (T) | Nerandomilast fed state (Test (T))/Nerandomilast fasted state (Reference (R))
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Washout period
Arm/Group | Nerandomilast fasted state (Reference (R))/Nerandomilast fed state Test (T) | Nerandomilast fed state (Test (T))/Nerandomilast fasted state (Reference (R))
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Nerandomilast fasted state (Reference (R))/Nerandomilast fed state Test (T) | Nerandomilast fed state (Test (T))/Nerandomilast fasted state (Reference (R))
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set includes all participants who were treated with at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nerandomilast Fasted State (Reference (R))/Nerandomilast Fed State Test (T) | Nerandomilast Fed State (Test (T))/Nerandomilast Fasted State (Reference (R)) | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] — Treated set (TS): The treated set includes all participants who were treated with at least one dose of trial drug.
  Years | 41.0 (7.1) | 38.0 (6.5) | 39.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Treated set (TS): The treated set includes all participants who were treated with at least one dose of trial drug.
  Participants
    Female | 4 | 4 | 8
    Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Treated set (TS): The treated set includes all participants who were treated with at least one dose of trial drug.
  Participants
    Hispanic or Latino | 0 | 1 | 1
    Not Hispanic or Latino | 9 | 8 | 17
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Treated set (TS): The treated set includes all participants who were treated with at least one dose of trial drug.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 9 | 9 | 18
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Nerandomilast in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point) (AUC0-tz)
Description: Area under the concentration-time curve of Nerandomilast in plasma over the time interval from 0 to the last quantifiable data point is presented.
  Geometric least square mean (adjusted geometric mean) and geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. These quantities will then be back-transformed to the original scale to provide the point estimate and 90% confidence intervals (CIs) for each endpoint. This model will include effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment.
Time Frame: Within 3 hours before Nerandomilast administration and at 0:15, 0:30, 0:45, 1:00, 1:15, 1:30, 1:45, 2:00, 2:30, 3:00, 3:30, 4:00, 6:00, 8:00, 11:00, 12:00, 24:00, 34:00, 48:00, 58:00, 72:00, 96:00, 120:00, and 144:00 hours after administration.
Population: Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomol/Liter (h*nmol/L)
Groups:
- Nerandomilast fasted state (Reference (R)): Participants received one 18 mg Nerandomilast Formulation C2 film-coated tablet following an overnight fast of at least 10 hours.
- Nerandomilast fed state (Test (T)): Participants received One 18 mg Nerandomilast Formulation C2 film-coated tablet following a high fat/high calorie meal.
Arm/Group | Nerandomilast fasted state (Reference (R)) | Nerandomilast fed state (Test (T))
Number analyzed (Participants) | 18 | 18
hour*nanomol/Liter (h*nmol/L) | 2225.20 (NA) — Geometric standard error = 1.07 | 2563.65 (NA) — Geometric standard error = 1.07
Statistical Analysis 1: Comparison: Nerandomilast fasted state (Reference (R)) vs Nerandomilast fed state (Test (T)); Relative bioavailability of Nerandomilast administered in fed state (Test) compared with Nerandomilast administered in fasted state (Reference) was estimated by the ratios of the gMeans (Test/Reference). Their corresponding 2-sided 90% confidence intervals (CIs) were provided. This method corresponds to 2 one-sided t-test procedures, each at the 5% significance level; Test type: Other; Ratios of adjusted geometric means [%] = 115.21, 90% CI 2-sided [106.55 to 124.58] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 13.5

2. Primary Outcome: Maximum Measured Concentration of Nerandomilast in Plasma (Cmax)
Description: Maximum measured concentration of Nerandomilast in plasma (Cmax) is presented.
  Geometric least square mean (adjusted geometric mean) and geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. These quantities will then be back-transformed to the original scale to provide the point estimate and 90% confidence intervals (CIs) for each endpoint. This model will include effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomol/Liter (nmol/L)
Arm/Group | Nerandomilast fasted state (Reference (R)) | Nerandomilast fed state (Test (T))
Number analyzed (Participants) | 18 | 18
nanomol/Liter (nmol/L) | 412.88 (NA) — Geometric standard error = 1.10 | 354.35 (NA) — Geometric standard error = 1.10
Statistical Analysis 1: Comparison: Nerandomilast fasted state (Reference (R)) vs Nerandomilast fed state (Test (T)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratios of adjusted geometric means [%] = 85.82, 90% CI 2-sided [68.80 to 107.06] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 39.4

3. Secondary Outcome: Area Under the Concentration-time Curve of Nerandomilast in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of Nerandomilast in plasma over the time interval from 0 extrapolated to infinity is presented.
  Geometric least square mean (adjusted geometric mean) and geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. These quantities will then be back-transformed to the original scale to provide the point estimate and 90% confidence intervals (CIs) for each endpoint. This model will include effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomol/Liter (h*nmol/L)
Arm/Group | Nerandomilast fasted state (Reference (R)) | Nerandomilast fed state (Test (T))
Number analyzed (Participants) | 18 | 18
hour*nanomol/Liter (h*nmol/L) | 2240.58 (NA) — Geometric standard error = 1.07 | 2578.16 (NA) — Geometric standard error = 1.07
Statistical Analysis 1: Comparison: Nerandomilast fasted state (Reference (R)) vs Nerandomilast fed state (Test (T)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratios of adjusted geometric means [%] = 115.07, 90% CI 2-sided [106.38 to 124.46] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 13.5

ADVERSE EVENTS:
Time Frame: Adverse event collection period: up to 7 days from first Nerandomilast administration. All-cause mortality: up to 28 days from first Nerandomilast administration.
Description: Treated set (TS): The treated set includes all participants who were treated with at least one dose of trial drug.
Arm/Group | Nerandomilast fasted state (Reference (R)) | Nerandomilast fed state (Test (T))
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 8/18 | 7/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nerandomilast fasted state (Reference (R)) (N=18) | Nerandomilast fed state (Test (T)) (N=18)
Flatulence (Gastrointestinal disorders) | 1 | 0
Catheter site pain (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 5
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT06415045/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT06415045/SAP_001.pdf